CLINICAL TRIAL: NCT03774459
Title: A Phase 2, Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Efficacy of ANAVEX2-73 for Cognitive Impairment in Patients With Parkinson's Disease With Dementia
Brief Title: ANAVEX2-73 Study in Parkinson's Disease Dementia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anavex Life Sciences Corp. (Industry)
Collaborators: Anavex Germany GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANAVEX2-73-PDD-001
Record Dates: First submitted 2018-12-08; First posted 2018-12-13 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Parkinsons Disease With Dementia
MeSH Terms: interventions — tetrahydro-N, N-dimethyl-2,2-diphenyl-3-furanmethanamine hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High dose ANAVEX2-73 (Experimental): High dose ANAVEX2-73
  Interventions: Drug: High dose ANAVEX2-73
- Mid dose ANAVEX2-73 (Experimental): Mid dose ANAVEX2-73
  Interventions: Drug: Mid dose ANAVEX2-73
- Placebo oral capsule (Placebo Comparator): Placebo oral capsule
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: High dose ANAVEX2-73 — Active oral capsule
  Arms: High dose ANAVEX2-73
Drug: Mid dose ANAVEX2-73 — Active oral capsule
  Arms: Mid dose ANAVEX2-73
Drug: Placebo oral capsule — Placebo oral capsule
  Arms: Placebo oral capsule

SUMMARY:
A Phase 2, Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Efficacy of ANAVEX2-73 for Cognitive Impairment in Patients with Parkinson's Disease with Dementia (PDD)

DETAILED DESCRIPTION:
This is a Phase 2, multicenter, randomized, double-blind, placebo-controlled, parallel-group, three-arm, 14-week study in PD patients with dementia. The study includes a 2 week Screening / Baseline Observation Period and a 14-week Treatment Period (including a 2 week Titration Period), and a 2-week Safety Follow-Up Period

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's disease (PD) consistent with the UK Parkinson's Disease Society Brain Bank diagnostic criteria.
* Diagnosis of probable PD dementia (PDD) according to the Movement Disorder Society Task Force clinical diagnostic criteria.
* Montreal Cognitive Assessment (MoCA) score of 13 to 23, inclusive, at Screening.
* Male or female and aged ≥ 50 years.
* Caregivers and subjects (or legal representative) must understand and have signed approved informed consent.
* Caregivers and subjects (or legal representative) must be able to understand study requirements and be willing to follow instructions.
* Stable regimen of anti-Parkinson's disease medications (including levodopa, dopamine agonists, MAO-B inhibitors, or the COMT inhibitor entacapone), which has been stable for at least 4 weeks prior to Baseline.
* Treatment with cholinesterase inhibitor (rivastigmine, donepezil and galantamine (Exelon®, Aricept®, or Reminyl®) will be permitted, provided the dose has been stable for a minimum of 8 weeks prior to randomization.
* Subjects with history of depression on antidepressant medications will be allowed if depression is controlled and they have been on a stable daily dose of the antidepressant for ≥8 weeks before Baseline.
* Contraception:

  * Women of childbearing potential must use an acceptable method of contraception starting 4 weeks prior to study drug administration and for a minimum of 4 weeks after study completion. Otherwise, women must be postmenopausal (at least one year absence of vaginal bleeding or spotting) as confirmed by FSH greater than or equal to 40 mIU/mL or 40 IU/L or be surgically sterile.
  * Men with a potentially fertile partner must have had a vasectomy or be willing to use an acceptable method of contraception for the duration of the study and for 3 months after study drug discontinuation.

Exclusion Criteria:

* History of any significant neurologic or psychiatric disorder other than PD that can contribute to cognitive impairment.
* Any other condition or clinically significant abnormal findings like severe co-morbidities e.g. history of stroke, poor kidney or liver function on the physical or neurological examination, medical and psychiatric history, at screening or at baseline that, in the opinion of the Investigator, would make the subject unsuitable for the study.
* Potential symptomatic causes of cognitive impairment including but not limited to

  1. abnormal thyroid function test at screening (TSH)
  2. abnormal B12 level at screening
  3. MRI findings (by history) pointing to a potential symptomatic cause of cognitive dysfunction, including significant vascular changes, or communicating hydrocephalus.
* Treatment with memantine or amantadine. If appropriate the drugs can be discontinued for a minimum of 4 weeks prior to randomization.
* Use of over the counter (OTC) or prescription medication for sleep on 2 or more occasions per week (less than that is allowed).
* History of depression as measured by Beck Depression Inventory score >17 at screening.
* Treatment with any other investigational drug or device within 4 weeks prior to screening.
* Smoking > 1 pack of cigarettes per day (as assessed for the 4 weeks prior to screening).
* Women who are pregnant or lactating.
* Known allergy or sensitivity to ANAVEX2-73 or any of its components.
* Suicidal ideation on the Columbia Suicide Severity Rating Scale (C-SSRS) of type 4 or type 5, or any suicidal behavior, in the past 6 months. Type 4 indicates active suicidal ideation with some intent to act, without a specific plan. Type 5 indicates active suicidal ideation with a specific plan and intent.
* Use of centrally acting anticholinergic drugs during the 4 weeks before randomization.
* Medications used for overactive bladder will be allowed provided that the regimen has been stable 4 weeks prior to randomization.
* Treatment with any dopamine receptor blocking medications with the exception of low dose quetiapine (≤50 mg/day). Pimavanserin (≤34 mg/day) will be allowed.
* History of neurosurgical intervention (e.g., deep brain stimulation) for PD.
* Unpredictable motor fluctuations that would interfere with administering cognitive assessments in the ON state.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Cognitive Drug Research (CDR) Computerized Assessment System Continuity of Attention | 14 weeks
  Change from Baseline to End of Treatment in Continuity of Attention as measured by Cognitive Drug Research (CDR) Computerized Assessment System Continuity of Attention test
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 14 weeks
  Assess the safety and tolerability of ANAVEX2-73 compared to placebo

SECONDARY OUTCOMES:
MDS-UPDRS Part III Total Score (Motor Scores) | 14 weeks
  Change from baseline to End of Treatment as measured by MDS-UPDRS Part III Total Score (Motor Scores)
SDS-CL-25 | 14 weeks
  Incidence of sleep disorders symptoms (SDS-CL-25)

CONTACTS AND LOCATIONS:
Locations (25):
- Australia (2):
  - KaRa MINDS, Macquarie Park
  - Hammond Health, Malvern
- Spain (23):
  - Hospital Cruces Bilbao, Barakaldo
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Mutua Terrasa, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital Universitario Puerta del Mar, Cadiz
  - Hospital del Henares, Coslada
  - Hospital General Universitario de Elche, Elche
  - Hospital Arquitecto Marcide, Ferrol
  - Hospital Santa Caterina, Girona
  - Clinica Ruber Internacional, Madrid
  - Clínica Universidad de Navarra (CUN) - Sede Madrid- Servicio de Neurología -, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital de La Princesa, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Infanta Leónor, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital HM Puerta del Sur, Móstoles
  - Hospital Universitario Central de Asturias (HUCA), Oviedo
  - Clínica Universidad de Navarra (CUN), Pamplona
  - Hospital de Santiago de Compostela, Santiago de Compostela
  - Hospital Universitario Virgen del Rocío, Seville